CLINICAL TRIAL: NCT03371758
Title: Expression of LC3-I, LC3-II & Beclin 1 in Vitiligo and Healthy Control; Comparative Study
Brief Title: Expression of LC3-I, LC3-II & Beclin 1 in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, Principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Dermatology
Record Dates: First submitted 2017-12-05; First posted 2017-12-13 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Autophagy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitiligo patients (Experimental)
  Interventions: Other: skin biopsy
- healthy controls (Experimental)
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — Punch skin biopsy will be taken from the lesional and non-lesional skin of vitiligo patients as well as healthy skin of controls.

SUMMARY:
The exact mechanism of impairment of autophagy in vitiligo has not yet been determined.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with non-segmental vitiligo whether active or stable.

  * Age above 12 years.
  * Both sexes.

Exclusion Criteria:

* • Patients should not use any topical or systemic treatment at least 6 weeks before inclusion into the study.

  * Patients having other autoimmune disease, heart disease, liver disease, kidney disease, neurological disorder, cancer, active infection or any chronic disease.
  * Pregnancy or breast feeding for female patients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Expression of LC3-I, LC3-II & Beclin 1 in vitiligo patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Fathy Elmasry, Cairo, Egypt